CLINICAL TRIAL: NCT03830515
Title: Evaluation of microMend Device to Close Skin Wounds Associated With Repair of Lacerations
Brief Title: Evaluation of microMend Device to Close Lacerations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KitoTech Medical, Inc. (Industry)
Collaborators: Brown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KTM005
Record Dates: First submitted 2019-02-02; First posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Lacerations; Wounds
Keywords: Lacerations; Wounds
MeSH Terms: conditions — Lacerations; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: A single arm open label study testing the ability of microMend to close lacerations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Closure of lacerations with microMend (Experimental): Laceration closure with microMend
  Interventions: Device: microMend

INTERVENTIONS:
Device: microMend — Wound closure product consisting of tan array of tiny metal Microstaples affixed to adhesive backing. The device is the size and shape of a butterfly closure and intended for closure of skin wounds.
  Other Names: microMend Skin Closure Device

SUMMARY:
In this study, total of 20 subjects will have lacerations will be closed with microMend, which is an FDA-listed wound closure product. microMend is a wound closure device that is the size and shape of a butterfly bandage and incorporates tiny Microstaples into an adhesive backing. Assessments by practitioners and Subjects of microMend will be made at Days 0 10, and 3 months using a combination of questionnaires and photographs.

DETAILED DESCRIPTION:
This is an open-label, single-arm Phase 2 Study to evaluate closure of skin wounds associated with laceration repair using microMend devices. A maximum of 20 Subjects will be enrolled in the Study in order to have 15 Subjects with evaluations at Month 3 after wound closure. The primary intent is to assess the wound closure results with microMend closure at Month 3 after the wound closure procedure. Evaluations will also take place at Days 0 and 10 and 1 Month post-procedure to assess wound closure results. An Independent Plastic Surgeon who is not closing wounds in the study will assess the efficacy of wound closure at Day 10, Month 1, and Month 3. Assessment will also be made of the Subject's pain with applying microMend, time of wound closure, and opinions of the Providers and Subjects about microMend.

Screening data will be reviewed to determine Subject eligibility. Subjects who meet all inclusion criteria and none of the exclusion criteria will be entered into the Study. The Provider may elect to close additional wounds in subjects who have more than one wound that qualifies for the study.

In the Study, eligible Subjects will undergo the laceration repair procedure as is standard and customary for each Provider except for skin closure will be performed using microMend devices. If more than one device is needed, the devices are to be applied adjacent to one another along the entire length of the wound. microMend devices are to be applied immediately adjacent to one another with no more than 1 mm separating each adjacent device. (Note: Each device closes 1-1.5 cm of wound length.). In addition, devices should be applied such that they extend to or beyond the ends of the wound along its length.

A minimum of two (2) photographs will be taken of each wound both before and after the application of microMend devices on the day of the wound closure procedure (Day 0).

If a wound is under high tension and/or has a maximum gap of more than 1 cm between the wound edges, it should be closed with subcutaneous sutures before applying microMend devices. If this is not performed, the wound should not be closed with microMend and the Subject is not eligible for the study.

Standard surgical staples, sutures, tissue adhesives, SteriStrips or other bandages should not be used to close any portion of skin wounds closed with microMend devices.

Each wound should be free of significant tissue injury and bleeding, contain no foreign bodies, and should be clean and completely dry and free of hair before application of microMend.

No other wound closure products, such as tissue adhesives, bandages such as SteriStrips, staples, or sutures should be applied to the wound.

Solutions, ointments, creams, and other moist materials should be avoided during the time period when the microMend remains on the skin except those recommended by the Provider.

After application of the microMend devices, it is recommended that each wound be covered with a non-stick gauze dressing. (Note: contact of adhesive with microMend devices is strictly prohibited.) Subject contact with the wound site should be minimized after placement of the microMend devices and the dressing. All other activities associated with the laceration repair procedure should follow the standard procedure used by the Provider. The Provider will fill out a questionnaire about the wound closure procedure. The Subject will rate the level of pain associated with microMend application.

The microMend devices are to be removed at the return clinic visit on Day 10 (acceptable range: Days 7-12) by the Provider (Physician, Nurse Practitioner, Physician's Assistant, or other qualified health care provider). Photographs are to be obtained of each wound both before and after removal of all microMend devices. A minimum of two (2) photographs will be taken of each wound both before and after removal of microMend devices. The Subject will fill out a questionnaire providing an opinion of microMend.

Each Subject is to return to the clinic at one (1) month post-procedure (acceptable range: Days 25-40) to obtain photographs of each wound. A minimum of two (2) photographs will be taken at the 1-month clinic visit. Each Subject is to return to the clinic at three (3) months after wound closure (acceptable range: 11-15 weeks) to obtain photographs of each wound. A minimum of two (2) photographs will be taken at the 1-month clinic visit.

Photographs obtained on Day 0, Day 10, Month 1, and Month 3 will be assessed for wound closure results by an Independent Plastic Surgeon, who is not performing laceration repair or wound closure in the study. The wound closure will be rated as either Satisfactory or Unsatisfactory. The quality of the wound closure will further be rated as Excellent, Good, Fair, or Poor. For Subjects that have had more than one wound closed with microMend devices, each wound is to be assessed separately at Day 0, Day 10, Month 1, and Month 3.

Total duration of Subject participation will be approximately 4 months, including screening, treatment, and follow-up.

ELIGIBILITY:
Inclusion Criteria

* Subjects undergoing a laceration repair that would require sutures, staples, or tissue adhesives to close the skin wound
* Age equal to or greater than 18 years old
* Written informed consent obtained from Subject or Subject's legal representative and ability for Subject to comply with the requirements of the Study

Exclusion Criteria

* Wound on face
* Wound on flexor surfaces such as over joints
* Wound on digits (fingers or toes)
* Wound under high tension, which is not closed with subcutaneous sutures before application of microMend devices
* Wound that has a gap of more than 1 cm between the wound edges immediately prior to application of microMend devices
* Wound with jagged or irregular edges
* Wound with significant tissue injury
* Visual evidence of active infection, contaminated or devitalized tissue, or rash at laceration location
* Wound that contain a foreign body
* Wound site that contains tattoo or other identifiable features
* Subject with keloid(s)
* Medical disorder that, in the opinion of the Provider, could have a significant effect on wound healing
* Pregnancy
* Inability of Subject to carry out Subject instructions
* Subject lacks the capacity to consent
* Medication that, in the opinion of the Provider, could have a significant effect on wound healing
* Skin disorder, such as psoriasis, or current dermatitis or eczema at wound site
* History of keloids or scar hypertrophy
* Known bleeding diathesis
* Sensitivity or allergy to adhesives or medical tape
* Active infection in any part of the body
* Use of sutures or staples in addition to microMend to close the outermost skin layer
* Use of tissue adhesive or other adhesives directly over the wound

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04-20 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Wound closure results of skin wounds after healing | 3 months
  Assessment of photographs of wounds closed with microMend at Monthg 3 by independent physician with experience in assessing skin wounds.
Overall assessment of microMend by Provider at end of the wound closure procedure. | Day 0
  Questionnaire on opinion of Provider (Physician, PA, or Nurse Practitioner on usability and other characteristics of microMend
Time of wound closure. | ay 0
  Measurement of time in seconds to close wound with microMend devices.
Subject's assessment of microMend. | Day 0
  Measurement of pain upon placement of microMend using VAS scoring system
Subject's assessment of pain with application of microMend | Day 10
  Questionnaire regarding evaluation of microMend

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Beaudoin, MD, PhD, Principal Investigator — Department of Emergency Medicine, Walpert School of Medicine, Brown University; Gregory Jay, MD, PhD, Principal Investigator — Department of Emergency Medicine, Walpert School of Medicine, Brown University
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nizami T, Beaudoin F, Suner S, Aluisio A, Bhatt RA, Jay GD. Evaluation of microMend wound closure device in repairing skin lacerations. Emerg Med J. 2023 Aug;40(8):564-568. doi: 10.1136/emermed-2022-212667. Epub 2023 May 23. PMID 37220958